CLINICAL TRIAL: NCT03373903
Title: A Multicenter, Dose-finding Study to Determine if Oral BEZ235 Alone or in Combination With RAD001 Decreases the Incidence of Respiratory Tract Infections in Elderly Subjects
Brief Title: Dose Finding Study to Determine if BEZ235 Alone or in Combination With RAD001 Decreases the Incidence of Respiratory Tract Infections in the Elderly
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Restorbio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RTB-BEZ235-202
Record Dates: First submitted 2017-11-20; First posted 2017-12-14 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections | interventions — dactolisib; Everolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo once daily for 16 weeks (Placebo Comparator)
  Interventions: Other: Placebo
- BEZ235 once daily for 16 weeks (Experimental)
  Interventions: Drug: BEZ235
- BEZ235 twice daily for 16 weeks (Experimental)
  Interventions: Drug: BEZ235
- BEZ235 plus RAD001 once daily for 16 weeks (Experimental)
  Interventions: Drug: BEZ235 plus everolimus (RAD001)

INTERVENTIONS:
Other: Placebo — oral
  Arms: Placebo once daily for 16 weeks
Drug: BEZ235 — oral
  Arms: BEZ235 once daily for 16 weeks; BEZ235 twice daily for 16 weeks
Drug: BEZ235 plus everolimus (RAD001) — Oral
  Arms: BEZ235 plus RAD001 once daily for 16 weeks

SUMMARY:
The purpose of this study is to evaluate the efficacy, tolerability, and safety of BEZ235 alone and in combination with RAD001 to support further development to reduce the incidence of respiratory tract infections (RTIs) in elderly subjects.

DETAILED DESCRIPTION:
This is a randomized, blinded, placebo-controlled, multicenter, parallel-group, dose finding 24-week study to assess the safety, tolerability and efficacy of up to 3 doses of BEZ235 alone and in combination with RAD001 as compared to placebo in elderly subjects who are at increased risk of respiratory tract infection related-morbidity and mortality. The study will be composed of up to a 6-week screening and run-in period, a 16-week treatment period and an 8-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects
* Age ≥ 85 years
* Age ≥ 65 and < 85 years with one or more of the following conditions:

  * Asthma
  * Chronic Obstructive Pulmonary Disease (COPD)
  * Chronic bronchitis
  * Type 2 Diabetes Mellitus (T2DM)
  * Congestive Heart Failure (CHF) New York Heart Association (NYHA) functional classification I-II
  * Current smoker
  * One or more emergency room visits or hospitalizations for a RTI during the previous 12 months

Exclusion Criteria:

* Subjects with medically significant cardiac conditions including NYHA functional classification III-IV
* Subjects with Type I diabetes mellitus.
* Subjects with clinically significant underlying pulmonary disease other than asthma, GOLD Class I and II COPD or chronic bronchitis
* History of malignancy in any organ system within the past 5 years except for the following:

  * Localized basal cell or squamous cell carcinoma of the skin, prostate cancer confined to the gland, cervical carcinoma in situ, breast cancer localized to the breast.
* Subjects with any one of the following:

  * hemoglobin < 10.0 g/dL for males and < 9.0 for females
  * white blood cell (WBC) count < 3,500/mm3,
  * neutrophil count < 2,000/mm3
  * platelet count < 125,000/mm3
* Subjects with a history of a systemic autoimmune disease or receiving immunosuppressive therapy
* Recent surgery other than minor skin surgery
* Liver disease or liver injury
* History or presence of impaired renal function
* History of immunodeficiency diseases
* Subjects with active infection
* Subjects with a Mini Mental Status Examination (MMSE) score <24 at screening.
* Significant illness (based on the subject's medical history and the clinical judgement of the investigator) which has not resolved within two (2) weeks prior to initial dosing.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 652 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
The percentage of subjects with 1 or more laboratory-confirmed RTIs through Week 16 | 16 weeks

SECONDARY OUTCOMES:
Percent of subjects who develop one or more RTIs through week 16 | 16 weeks
The rate of RTIs/person through week 16 | 16 weeks
The rate of RTIs per person through week 24 | 24 weeks
The percentage of subjects with 1 or more laboratory-confirmed RTIs through week 24 | 24 weeks
Peak Plasma Concentration (Cmax) | 8 weeks
Area under the plasma concentration versus time curve (AUC) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sarb Shergill, PhD, Study Director — Restorbio Inc.
Locations (1):
- Heartland Research Associates, Wichita, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mannick JB, Teo G, Bernardo P, Quinn D, Russell K, Klickstein L, Marshall W, Shergill S. Targeting the biology of ageing with mTOR inhibitors to improve immune function in older adults: phase 2b and phase 3 randomised trials. Lancet Healthy Longev. 2021 May;2(5):e250-e262. doi: 10.1016/S2666-7568(21)00062-3. Epub 2021 May 6. PMID 33977284